CLINICAL TRIAL: NCT01087996
Title: A Phase I/II, Randomized Pilot Study of the Comparative Safety and Efficacy of Transendocardial Injection of Autologous Mesenchymal Stem Cells Versus Allogeneic Mesenchymal Stem Cells in Patients With Chronic Ischemic Left Ventricular Dysfunction Secondary to Myocardial Infarction
Brief Title: The Percutaneous Stem Cell Injection Delivery Effects on Neomyogenesis Pilot Study (The POSEIDON-Pilot Study)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Joshua M Hare, Director, Interdisciplinary Stem Cell Institute, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20090352; R01HL110737 (NIH); R01HL107110 (NIH); R01HL084275 (NIH); P20HL101443 (NIH); R01HL094849 (NIH)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Stem Cell Transplantation
Keywords: Chronic Ischemic Left Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Auto-hMSCs (Experimental): Participants will receive an injection of 20 million, 100 million or 200 million autologous human mesenchymal stem cells.
  Interventions: Biological: Auto-hMSCs
- Allo-hMSCs (Experimental): Participants will receive an injection of 20 million, 100 million or 200 million allogeneic human mesenchymal stem cells.
  Interventions: Biological: Allo-hMSCs

INTERVENTIONS:
Biological: Auto-hMSCs — Biological: Autologous human mesenchymal stem cells (Auto-hMSCs) Participants will receive 40 million cells/mL delivered in either a dose of 0.5 mL per injection x 1 injection for a total of 0.2 x 10^8 (20 million) Auto-hMSCs, a dose of 0.5 mL per injection x 5 injections for a total of 1 x 10^8 (100 million) Auto-hMSCs, or a dose of 0.5 mL per injection x 10 injections for a total of 2 x 10^8 (200 million) Auto-hMSCs. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
  Arms: Auto-hMSCs
Biological: Allo-hMSCs — Biological: Allogeneic human mesenchymal stem cells (Allo-hMSCs) Participants will receive 40 million cells/mL delivered in either a dose of 0.5 mL per injection x 1 injection for a total of 0.2 x 10^8 (20 million) Allo-hMSCs, a dose of 0.5 mL per injection x 5 injections for a total of 1 x 10^8 (100 million) Allo-hMSCs, or a dose of 0.5 mL per injection x 10 injections for a total of 2 x 10^8 (200 million) Allo-hMSCs. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
  Arms: Allo-hMSCs

SUMMARY:
The technique of transplanting progenitor cells into a region of damaged myocardium, termed cellular cardiomyoplasty, is a potentially new therapeutic modality designed to replace or repair necrotic, scarred, or dysfunctional myocardium. Ideally, graft cells should be readily available, easy to culture to ensure adequate quantities for transplantation, and able to survive in host myocardium; often a hostile environment of limited blood supply and immunorejection. Whether effective cellular regenerative strategies require that administered cells differentiate into adult cardiomyocytes and couple electromechanically with the surrounding myocardium is increasingly controversial, and recent evidence suggests that this may not be required for effective cardiac repair. Most importantly, transplantation of graft cells should improve cardiac function and prevent adverse ventricular remodeling. To date, a number of candidate cells have been transplanted in experimental models, including fetal and neonatal cardiomyocytes, embryonic stem cell-derived myocytes, tissue engineered contractile grafts, skeletal myoblasts, several cell types derived from adult bone marrow, and cardiac precursors residing within the heart itself. There has been substantial clinical development in the use of whole bone marrow and skeletal myoblast preparations in studies enrolling both post-infarction patients, and patients with chronic ischemic left ventricular dysfunction and heart failure. The effects of bone-marrow derived mesenchymal stem cells (MSCs) have also been studied clinically.

Currently, bone marrow or bone marrow-derived cells represent highly promising modality for cardiac repair. The totality of evidence from trials investigating autologous whole bone marrow infusions into patients following myocardial infarction supports the safety of this approach. In terms of efficacy, increases in ejection fraction are reported in the majority of the trials.

Chronic ischemic left ventricular dysfunction resulting from heart disease is a common and problematic condition; definitive therapy in the form of heart transplantation is available to only a tiny minority of eligible patients. Cellular cardiomyoplasty for chronic heart failure has been studied less than for acute MI, but represents a potentially important alternative for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic ischemic left ventricular dysfunction secondary to MI.
* Be a candidate for cardiac catheterization.
* Been treated with appropriate maximal medical therapy for heart failure or post-infarction left ventricular dysfunction.
* Ejection fraction between 20% and 50%.
* Able to perform a metabolic stress test.

Exclusion Criteria:

* Baseline glomerular filtration rate <50 ml/min/1.73m2.
* Presence of a mechanical aortic valve or heart constrictive device.
* Documented presence of aortic stenosis (aortic stenosis graded as ≥+2 equivalent to an orifice area of 1.5cm2 or less).
* Documented presence of moderate to severe aortic insufficiency (echocardio- graphic assessment of aortic insufficiency graded as ≥+2).
* Evidence of a life-threatening arrhythmia (nonsustained ventricular tachycardia ≥20 consecutive beats or complete heart block) or QTc interval >550 ms on screening ECG. In addition; patients with sustained or a short run of ventricular tachycardia on ECG or 48 hour Ambulatory ECG during the screening period will be removed from the protocol.
* Documented unstable angina.
* AICD firing in the past 60 days prior to the procedure.
* Be eligible for or require coronary artery revascularization.
* Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet values < 100,000/ul without another explanation.
* Have liver dysfunction, as evidenced by enzymes (ALT and AST) greater than three times the ULN.
* Have a coagulopathy condition = (INR > 1.3) not due to a reversible cause.
* Known, serious radiographic contrast allergy.
* Known allergies to penicillin or streptomycin.
* Organ transplant recipient.
* Clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
* Non-cardiac condition that limits lifespan to < 1 year.
* On chronic therapy with immunosuppressant medication.
* Serum positive for HIV, hepatitis BsAg, or hepatitis C.
* Female patient who is pregnant, nursing, or of child-bearing potential and not using effective birth control.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Result] Hare JM, Fishman JE, Gerstenblith G, DiFede Velazquez DL, Zambrano JP, Suncion VY, Tracy M, Ghersin E, Johnston PV, Brinker JA, Breton E, Davis-Sproul J, Schulman IH, Byrnes J, Mendizabal AM, Lowery MH, Rouy D, Altman P, Wong Po Foo C, Ruiz P, Amador A, Da Silva J, McNiece IK, Heldman AW, George R, Lardo A. Comparison of allogeneic vs autologous bone marrow-derived mesenchymal stem cells delivered by transendocardial injection in patients with ischemic cardiomyopathy: the POSEIDON randomized trial. JAMA. 2012 Dec 12;308(22):2369-79. doi: 10.1001/jama.2012.25321. PMID 23117550
- [Derived] Tompkins BA, Rieger AC, Florea V, Banerjee MN, Natsumeda M, Nigh ED, Landin AM, Rodriguez GM, Hatzistergos KE, Schulman IH, Hare JM. Comparison of Mesenchymal Stem Cell Efficacy in Ischemic Versus Nonischemic Dilated Cardiomyopathy. J Am Heart Assoc. 2018 Jul 12;7(14):e008460. doi: 10.1161/JAHA.117.008460. PMID 30005555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between April 2, 2010 and September 14, 2011
Pre-assignment Details: One patient did not receive Autologous MSCs because they became ineligible.
Groups:
- Allo-hMSCs: Participants will receive an injection of 20 million, 100 million or 200 million allogeneic human mesenchymal stem cells.
  Allo-hMSCs : Biological: Allogeneic human mesenchymal stem cells (Allo-hMSCs) Participants will receive 40 million cells/mL delivered in either a dose of 0.5 mL per injection x 1 injection for a total of 0.2 x 10^8 (20 million) Allo-hMSCs, a dose of 0.5 mL per injection x 5 injections for a total of 1 x 10^8 (100 million) Allo-hMSCs, or a dose of 0.5 mL per injection x 10 injections for a total of 2 x 10^8 (200 million) Allo-hMSCs. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
- Auto-hMSCs: Participants will receive an injection of 20 million, 100 million or 200 million autologous human mesenchymal stem cells.
  Auto-hMSCs : Biological: Autologous human mesenchymal stem cells (Auto-hMSCs) Participants will receive 40 million cells/mL delivered in either a dose of 0.5 mL per injection x 1 injection for a total of 0.2 x 10^8 (20 million) Auto-hMSCs, a dose of 0.5 mL per injection x 5 injections for a total of 1 x 10^8 (100 million) Auto-hMSCs, or a dose of 0.5 mL per injection x 10 injections for a total of 2 x 10^8 (200 million) Auto-hMSCs. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
Period: Overall Study
Arm/Group | Allo-hMSCs | Auto-hMSCs
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allo-hMSCs | Auto-hMSCs | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.5) | 63.7 (9.3) | 63.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Incidence of TE-SAE Define as Composite of Death, Non-fatal MI, Stroke, Hospitalization for Worsening Heart Failure, Cardiac Perforation, Pericardial Tamponade, Ventricular Arrhythmias >15 Sec. or With Hemodynamic Compromise or Atrial Fibrillation
Time Frame: One month post-catheterization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 15 | 15
percentage of participants | 6.70 [1.70 to 31.95] | 6.70 [1.70 to 31.95]
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p = 1.00, Fisher Exact

2. Secondary Outcome: CT Infarct Size From Early Enhanced Defect: - Difference Between the Baseline and 13-month
Description: Percentage change from 13-months post-catheterization to baseline.
Time Frame: Baseline Month 13 post-catheterization
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 15 | 15
percent change from baseline | -31.61 [-49.24 to -13.99] | -34.93 [-48.18 to -21.68]
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p = 0.75, ANOVA

3. Secondary Outcome: CT Measure of Left Ventricular Ejection Fraction
Time Frame: Baseline Month 13 post-catheterization
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 15 | 15
percent
  Baseline | 27.85 [22.30 to 33.41] | 26.23 [20.26 to 32.20]
  13-Month | 29.50 [24.10 to 34.90] | 28.53 [23.40 to 33.66]
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: CT Measure of End Diastolic Volume
Time Frame: Baseline Month 13 post-catheterization
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 15 | 15
ml
  Baseline | 260.26 [211.21 to 309.31] | 300.89 [251.33 to 350.45]
  13-Month | 243.66 [200.17 to 287.14] | 291.75 [235.45 to 348.05]
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p > 0.05, ANOVA

5. Secondary Outcome: CT Measure of End Systolic Volume
Time Frame: Baseline Month 13 post-catheterization
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 15 | 15
ml
  Baseline | 191.95 [145.77 to 238.12] | 225.67 [178.46 to 272.88]
  13-Month | 175.99 [135.21 to 216.46] | 213.59 [164.26 to 262.93]
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p > 0.05, ANOVA

6. Secondary Outcome: CT Measure of Scar Size as % of LV Mass
Time Frame: Baseline Month 13 post-catheterization
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 15 | 15
percent
  Baseline | 9.40 [7.11 to 11.68] | 10.71 [6.99 to 14.43]
  Month 13 | 5.54 [3.92 to 7.16] | 5.92 [4.16 to 7.67]
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p > 0.05, ANOVA

7. Secondary Outcome: Change in Distance Walked in 6-minutes From Baseline.
Time Frame: 12-months
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 15 | 15
meters | 19.7 [-19.0 to 58.3] | 65.8 [27.2 to 104.5]
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p = 0.87, Repeated measures ANOVA

8. Secondary Outcome: Change in Minnesota Living With Heart Failure Total Score
Description: The Minnesota living with heart failure questionnaire uses a 6-point, zero to five, Likert scale. The total score is the sum of the 21 responses. The total score is considered the best measure of how heart failure and treatments impact a patients quality of life. The max score is 105, minimum score is 0. A lower score is considered a better quality of life.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 15 | 15
units on a scale | -10.2 [-31.1 to 10.7] | -13.0 [-22.6 to -3.3]
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p = 0.84, Repeated measures ANOVA

9. Secondary Outcome: Change in New York Heart Association Class at 12-months
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Allo-hMSCs | Auto-hMSCs
Number analyzed (Participants) | 14 | 14
participants
  Improved NYHA Class | 4 | 7
  No change in NYHA Class | 8 | 6
  Worsened NYHA Class | 2 | 1
Statistical Analysis 1: Comparison: Allo-hMSCs vs Auto-hMSCs; Test type: Superiority or Other; p = 0.55, Chi-squared

ADVERSE EVENTS:
Description: Adverse events are shown by organ system.
Arm/Group | Allo-hMSCs | Auto-hMSCs
Serious Adverse Events (participants affected / at risk) | 5/15 | 8/15
Other Adverse Events (participants affected / at risk) | 10/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allo-hMSCs (N=15) | Auto-hMSCs (N=15)
Cardiac Disorders (Cardiac disorders) | 3 (3) | 7 (7)
Nervous System Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Renal and Urinary Disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory, Thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1) | 0 (0)
Surgical and Medical Procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Vascular Disorders (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allo-hMSCs (N=15) | Auto-hMSCs (N=15)
cardiac disorder (Cardiac disorders) | 6 (6) | 7 (7)
Eye Disorders (Eye disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 3 (3)
General disorders and administration site conditions (General disorders) | 1 (1) | 2 (2)
Infections and infestations (Infections and infestations) | 3 (3) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Musculoskeletal and connective issue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Nervous System Disorders (Nervous system disorders) | 0 (0) | 4 (4)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Skin and subcutaneous disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
vascular disorders (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No